CLINICAL TRIAL: NCT04078802
Title: Transvaginal Natural Orifice Transluminal Endoscopic Surgery (vNOTES) Compared With Traditional Vaginal Utero-sacral Ligament Suspension for Vaginal Apex Prolapse
Brief Title: 0050-19-RMB CTIL - VNOTES Compared to VH for Vaginal Apex Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, Omer MOR MD, Principle Investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RambamMD
Record Dates: First submitted 2019-09-02; First posted 2019-09-06 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Vaginal Prolapse
MeSH Terms: conditions — Uterine Prolapse

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VNOTES ARM (Experimental): treatment of Vaginal prolapse with VNOTES surgery and apical suspension to the uterosacral ligaments.
  Interventions: Procedure: VNOTES/VH
- Vaginal hysterectomy Arm (Experimental): treatment of Vaginal prolapse with classic vaginal hysterectomy surgery and apical suspension to the uterosacral ligaments.
  Interventions: Procedure: VNOTES/VH

INTERVENTIONS:
Procedure: VNOTES/VH — same as above

SUMMARY:
VNOTES (Transvaginal natural orifice transluminal endoscopic surgery) is a relatively new surgery for Hysterectomy and Uterosacral ligament suspension to treat Vaginal prolapse. The investigators wish to run a randomized control trial comparing it to classic Vaginal hysterectomy for the same indication.

DETAILED DESCRIPTION:
The investigators will recruit 60 women with indication for surgery to treat uterine prolapse. 30 women will undergo VNOTES surgery and 30 women will undergo classic vaginal hysterectomy. The investigators will compare outcomes of the surgeries such as surgery time, bleeding and clinical outcomes after 3 and 6 months post operation.

ELIGIBILITY:
Inclusion Criteria:

* women with vaginal prolapse
* capable of having a surgery - assessed by an anesthesiologist
* women who approve of having the surgery

Exclusion Criteria:

* BMI over 40
* women who have recurrent PID (pelvic inflammatory disease)
* women with oncology records

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only women suffer from vaginal prolapse
Enrollment: 60 (Estimated)
Dates: Start 2019-10 (Estimated); Primary Completion 2020-10 (Estimated); Study Completion 2020-11 (Estimated)

PRIMARY OUTCOMES:
surgery time | from admission up to 6 hours post operation
  time of surgery

SECONDARY OUTCOMES:
bleeding | from admission up to 6 hours post operation
  bleeding at surgery - volume of blood loss estimated by the surgeon performing the operation.
hospital days | from admission up to 96 hours post operation
  how many days after surgery for hospitalization
PISQ12 score - Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire | from admission up to 6 hours post operation
  Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire is a scoring index used to measure sexual function of women affected by pelvic organ prolapse. range 0-48. 0 marks good sexual function and 48 measures sexual disability affected from pelvic organ prolapse
PFDI score - Pelvic Floor Disability Index | from admission up to 6 hours post operation
  The Pelvic Floor Disability Index is an index used to obtain an objective score regarding pelvic floor disability comprising of bowel, bladder, or pelvic symptoms over the last 3 months prior to answering the questionnaire. score ranges 0-300. 0 outcome is no pelvic floor disability and 300 marks a high level of pelvic floor disability.

CONTACTS AND LOCATIONS:
Overall Officials: Omer Mor, MD, Principal Investigator — Rambam Health Care Campus

IPD SHARING:
Plan to Share IPD: No